CLINICAL TRIAL: NCT07266883
Title: Targeting the Brain-gut Axis in Inflammatory Bowel Diseases: Implementation and Exploration of Mechanism and Early Effectiveness of a Mindfulness-based Stress Reduction Program
Brief Title: A Mindfulness-based Stress Reduction Program for IBD
Acronym: MBSRforIBD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 75285
Record Dates: First submitted 2025-09-10; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-09

CONDITIONS: Inflammatory Bowel Disease (Crohn&Amp;#39;s Disease and Ulcerative Colitis)
Keywords: IBD; psychological distress; mindfulness
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBSR group (Experimental): Will participate in an 8 week mindfulness based stress reduction course, administered by a trained professional (clinician), virtually (zoom) with sessions once weekly and homework exercises. Group format.
  Interventions: Behavioral: Mindfulness based stress reduction
- Active Control (Active Comparator): Will be asked to watch an educational video on stress reduction
  Interventions: Other: Active Control

INTERVENTIONS:
Behavioral: Mindfulness based stress reduction — Mindfulness based stress reduction (MBSR) course. Participants will complete this course, which will have weekly sessions over Zoom (group format) over 8 weeks. Homework exercises will also be part of the course.
  Arms: MBSR group
Other: Active Control — Educational stress reduction video
  Arms: Active Control

SUMMARY:
The gut-brain connection is important for good health and when it is disrupted it can worsen existing chronic disease. Studies have shown that chronic stress has negative effects on the gastrointestinal tract such as inflammation and disruption of the beneficial bacteria that live there. These negative effects of chronic stress can lead to flare-ups of IBD. Mindfulness-based stress reduction (MBSR) is a structured 8 week program that aims to reduce stress by teaching mindfulness techniques. Recent research in people living with IBD suggest that MBSR could improve their quality of life by reducing stress levels.

The study aims to investigate the effects of MBSR on both the mental health of people living with IBD, and their physical health. We are studying people who are participating in an MBSR program as well as those receiving standard care at the QEII Health Sciences Centre. This study will assess how effective the MBSR program is compared to standard care at reducing distress and signs of stress and inflammation in people living with IBD. This study hopes to provide valuable insights into how mindfulness techniques could be used to support individuals living with IBD. Ultimately, this research aims to improve quality of life and health outcomes for people affected by this challenging condition.

DETAILED DESCRIPTION:
Inflammatory bowel diseases (IBD), including Crohn's disease (CD) and ulcerative colitis (UC), are chronic immune-mediated diseases that affect the gastrointestinal tract most often diagnosed in the second and third decades of life. IBD can have a deleterious impact on one's personal life, work and career trajectory, and mental and physical health over time. Untreated, IBD often leads to significant impairments in quality of life related to the effect of the disease on both mental and physical health . More than 30 percent of people living with IBD are also struggling with some form of psychological distress (PD) at any given time, which may be a result of the disease or independent of IBD. Forms of PD include, but are not limited to, anxiety, depression, and disease-related stress. .

Although psychotherapy interventions have been the main focus for management of psychological distress in IBD, a growing body of literature focusing on mindfulness based interventions (MBIs) in IBD exists . MBI interventions center around the development of greater capacity for "awareness that arises through paying attention, on purpose, in the present moment, non-judgementally". Greater capacity to default to present moment awareness rather than a future focus, specifically, excessive worrying (fuels anxiety) or backward gazing, specifically ruminating (predisposes to depression) has the potential to significantly improve chronic disease-related distress in persons living with IBD. One of the most well-defined, evidence-based MBIs is a structured, standardized, 8-week curriculum centered on experiential learning and mindfulness practices called mindfulness-based stress reduction the promise of MBSR, many questions remain unanswered. Variability in IBD patient populations studied, nature and severity of psychological distress, outcome measures, study design, and overall lack of mechanistic research in IBD are all gaps in existing research that need to be addressed. The benefit of MBSR to target the brain-gut axis and as an adjunctive therapy is also unclear.

The Nova Scotia collaborative IBD program is running an 8-week MBSR program for people in N.S. living with IBD. With this prospective observational cohort study, we plan to evaluate how effective this program is in improving quality of life and reducing stress biomarkers and psychological stress scores for adult patients with IBD. This study will compare health outcomes of patients who participated in an MBSR program run by qualified MBSR teachers affiliated with the NSCIBD to a group of patients who've received standard of care.

The overall objectives of this study are to:

1. Evaluate the early effectiveness of the 8-week MBSR program and
2. Collect and analyze biological and microbial markers of systemic and intestinal inflammation to understand MBSR-mediated psychological, disease-related, immunologic, neurohormonal, and microbiome impacts in persons living with mild to moderately active IBD compared to controls.

This will be an open label, comparator controlled study in which patients with IBD will undergo random allocation to either standard of care + a stress reduction education educational video or standard care + an 8 week MBSR program (MBSR-IBD). MBSR is skills-based, experiential learning program in which participants attend weekly 2.5 hour sessions for 8 weeks plus one full day weekend session. Over the course of these sessions participants learn mindfulness-based skills including, but not limited to, formal and informal meditation. Inclusion criteria include participants 18 years of age or older, having a known diagnosis of IBD that is mildly to moderately active. Health outcome data on clinical disease activity, microbial diversity, and cytokine arrays will be prospectively collected. Psychological questionnaires will also be collected. Data on disease activity, duration, phenotype, as well as medication and surgical history will be collected via targeted chart review.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* having a known diagnosis of IBD that is mildly to moderately active

Exclusion Criteria:

* pediatric participants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Psychological distress (GAD7) | Visit 1 (2 months post enrollment)
  Participant psychological distress, measured by the Generalized Anxiety Disorder Assessment (GAD7) scale
Psychological distress (GAD7) | Visit 2 (6 months post enrollment)
  Participant psychological distress, measured by the Generalized Anxiety Disorder Assessment (GAD7) scale
Psychological distress (PHQ9) | Visit 1 (2 months post enrollment)
  Participant psychological distress, measured by the eight-item Patient Health Questionnaire depression (PHQ9) scale
Psychological distress (PHQ9) | Visit 2 (6 months post enrollment)
  Participant psychological distress, measured by the eight-item Patient Health Questionnaire depression (PHQ9) scale
IBD Related quality of life score (SIBDQ) | Visit 1 (2 months post enrollment)
  IBD Related quality of life score, measured by the Short Inflammatory Bowel Disease Questionnaire (SIBDQ)
IBD Related quality of life score (SIBDQ) | Visit 2 (6 months post enrollment)
  IBD Related quality of life score, measured by the Short Inflammatory Bowel Disease Questionnaire (SIBDQ)
General quality of life score (SF-36) | Visit 1 (2 months post enrollment)
  General quality of life score, measured by the SF-36 questionnaire
General quality of life score (SF-36) | Visit 2 (6 months post enrollment)
  General quality of life score, measured by the SF-36 questionnaire

SECONDARY OUTCOMES:
Mindfulness (FFMQ) | Visit 1 (2 months post enrollment)
  Participant mindfulness, measured by the Five Facet Mindfulness Questionnaire (FFMQ)
Mindfulness (FFMQ) | Visit 2 (6 months post enrollment)
  Participant mindfulness, measured by the Five Facet Mindfulness Questionnaire (FFMQ)
Resilience (CD-RISC) | Visit 1 (2 months post enrollment)
  Participant psychological resilience, measured by the Connor-Davidson Resilience Scale (CD-RISC)
Resilience (CD-RISC) | Visit 2 (6 months post enrollment)
  Participant psychological resilience, measured by the Connor-Davidson Resilience Scale (CD-RISC)
Participant Self efficacy score (NGSE Scale) | Visit 1 (2 months post enrollment)
  Self-efficacy, measured by the New General Self Efficacy Scale
Participant Self efficacy score (NGSE Scale) | Visit 2 (6 months post enrollment)
  Self-efficacy, measured by the New General Self Efficacy Scale (NGSE Scale)
Psychological Flexibility (compACT) | Visit 1 (2 months post enrollment)
  Participant psychological flexibility, measured by the Comprehensive assessment of Acceptance and Commitment Therapy processes (CompACT) scale
Psychological Flexibility (compACT) | Visit 2 (6 months post enrollment)
  Participant psychological flexibility, measured by the Comprehensive assessment of Acceptance and Commitment Therapy processes (CompACT) scale
Participant Fatigue (FACIT-F) | Visit 1 (2 months post enrollment)
  Participant fatigue as measured by the Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) Scale
Participant Fatigue (FACIT-F) | Visit 2 (6 months post enrollment)
  Participant fatigue as measured by the Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) Scale
Fecal microbial diversity | Visit 1 (8 weeks post enrollment)
  Participant fecal microbial diversity, measured as laboratory based estimates of alpha diversity, beta-diversity, from processed fecal samples.
Fecal microbial diversity | Visit 2 (6 months post enrollment)
  Participant fecal microbial diversity, measured as laboratory based estimates of alpha diversity, beta-diversity, from processed fecal samples.
Fecal microbial abundance | Visit 1 (2 months post enrollment)
  Participant fecal microbial abundance, measured as laboratory based estimates of relative abundance of individual amplicon sequence variants (ASVs)from processed fecal samples.
Fecal microbial abundance | Visit 2 (6 months post enrollment)
  Participant fecal microbial abundance, measured as laboratory based estimates of relative abundance of individual amplicon sequence variants (ASVs)from processed fecal samples.

CONTACTS AND LOCATIONS:
Locations (1):
- QEII Health Sciences Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: Undecided